CLINICAL TRIAL: NCT04225845
Title: The Economic Consequences of Loneliness Among the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Abdul Latif Jameel Poverty Action Lab (Other)
Responsible Party: Principal Investigator, Esther Duflo, Research Associate, NBER; Abdul Latif Jameel Professor of Poverty Alleviation and Development Economics, MIT, National Bureau of Economic Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 172020; P01AG005842 (NIH)
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phone therapy (Experimental): Weekly phone calls by lay trained personnel to deliver problem solving therapy.
  Interventions: Behavioral: Phone therapy
- Phone therapy plus cash transfer (Experimental): Weekly phone calls by lay trained personnel to deliver problem solving therapy. Combined with a one-time cash transfer of Rs.1000.
  Interventions: Behavioral: Phone therapy; Behavioral: Cash transfer
- Cash transfer (Experimental): One-time cash transfer of Rs.1000.
  Interventions: Behavioral: Cash transfer
- Control (No Intervention): Control group.

INTERVENTIONS:
Behavioral: Phone therapy — Weekly phone calls by lay trained personnel to deliver problem solving therapy.
  Arms: Phone therapy; Phone therapy plus cash transfer
Behavioral: Cash transfer — One-time cash transfer of Rs.1000.
  Arms: Cash transfer; Phone therapy plus cash transfer

SUMMARY:
Elderly individuals across the world are increasingly living alone. However, little is known about the effects of loneliness on economic and health outcomes. The elderly living alone (i.e., in a household of size 1) will be randomized into one of two cross-randomized intervention arms or a control condition to improve older individuals' mental wellbeing as well as ability to cover basic needs, particularly in times of COVID (including health). The first intervention will focus on improving the elderly's outlook on life and relationships through problem-solving therapy (PST) delivered over the phone. The second will deliver to them a one-time cash transfer of Rs.1000, equivalent to the emergency help amount distributed to ration card holder by the government of Tamil Nadu. Each intervention will be offered on its own in each of two treatment arms, and in combination in a third. A control group will receive no intervention. Investigators will track outcomes of the elderly at 3 weeks and 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 55 years of age
* Individuals living alone

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1120 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Difficulty in performing daily activities/Functional impairment score | Assessed at 3 weeks after intervention
  Participants will be asked the level of difficulty they have in doing each of the following tasks: standing for 30 minutes, walking a long distance (1km), concentrating for 10 minutes, learning a new task like getting to a new place, washing whole body, getting dressed, taking care of household activities, doing day-to-day work, dealing with people they do not know, maintaining a friendship, being emotionally affected by health problems, and joining in community activities. The scale is from 0-4, with 0 being no difficulty, 1 mild, 2 moderate, 3 severe, and 4 cannot do. The scores will be summed to create a cumulative score on a 0-48 scale.
Difficulty in performing daily activities/Functional impairment score | Assessed at 3 months after intervention
  Participants will be asked the level of difficulty they have in doing each of the following tasks: standing for 30 minutes, walking a long distance (1km), concentrating for 10 minutes, learning a new task like getting to a new place, washing whole body, getting dressed, taking care of household activities, doing day-to-day work, dealing with people they do not know, maintaining a friendship, being emotionally affected by health problems, and joining in community activities. The scale is from 0-4, with 0 being no difficulty, 1 mild, 2 moderate, 3 severe, and 4 cannot do. The scores will be summed to create a cumulative score on a 0-48 scale.
Mental health | Assessed at 3 weeks after intervention
  The geriatric depression index short form is used. Participants are asked yes/no questions: if they are satisfied with their lives, have dropped activities and interests, feel their life is empty, often get bored, in good spirits most of the time, afraid that something bad is going to happen to them, feel happy most of the time, often feel hopeless, prefer to stay at home, rather than going out and doing new things, have problems with memory, think it is wonderful to be alive, feel worthless, feel full of energy, feel lonely, feel their situation is hopeless, think that most people are better off than they are. Responses will be summed over these questions.
Mental health | Assessed at 3 months after intervention
  The geriatric depression index short form is used. Participants are asked yes/no questions: if they are satisfied with their lives, have dropped activities and interests, feel their life is empty, often get bored, in good spirits most of the time, afraid that something bad is going to happen to them, feel happy most of the time, often feel hopeless, prefer to stay at home, rather than going out and doing new things, have problems with memory, think it is wonderful to be alive, feel worthless, feel full of energy, feel lonely, feel their situation is hopeless, think that most people are better off than they are. Responses will be summed over these questions.
Food security | Assessed at 3 weeks after intervention
  Participants will be asked to report whether in the past week they had to skip or cut the size of meals in the past week.
Food security | Assessed at 3 months after intervention
  Participants will be asked to report whether in the past week they had to skip or cut the size of meals in the past week.

SECONDARY OUTCOMES:
Seeking or receiving COVID vaccine | Assessed at 3 weeks after intervention
  Participants will be asked if they received the COVID vaccine or sought it (went to the health center but there was no availability).
Seeking or receiving COVID vaccine | Assessed at 3 months after intervention
  Participants will be asked if they received the COVID vaccine or sought it (went to the health center but there was no availability).
Loneliness | Assessed at 3 weeks after intervention
  Measured using the short-form University of California, Los Angeles (UCLA) Loneliness Scale (aka ULS-4). This is a 4-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. The questions are: no one really knows me well, people are around me but not with me, I feel in tune with the people around me, I can find companionship when I want it. Subjects rate each item as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"). Responses are summed over the four questions and rescaled to a 0-1 scale.
Loneliness | Assessed at 3 months after intervention
  Measured using the short-form University of California, Los Angeles (UCLA) Loneliness Scale (aka ULS-4). This is a 4-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. The questions are: no one really knows me well, people are around me but not with me, I feel in tune with the people around me, I can find companionship when I want it. Subjects rate each item as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"). Responses are summed over the four questions and rescaled to a 0-1 scale.
Healthcare utilization | Assessed at 3 weeks after intervention
  Participants will be asked if they fell ill in the last week, and, if yes, whether they used a medical provider or pharmacy to deal with the illness (0/1).
Healthcare utilization | Assessed at 3 months after intervention
  Participants will be asked if they fell ill in the last week, and, if yes, whether they used a medical provider or pharmacy to deal with the illness (0/1).
Survival of elderly person | Assessed at 3 weeks after intervention
  Whether still living at time of follow-up survey (0/1 variable)
Survival of elderly person | Assessed at 3 months after intervention
  Whether still living at time of follow-up survey (0/1 variable)
Social integration: non-family | Assessed at 3 weeks after intervention
  This is an indicator for whether the participant talked on the phone with anyone (with the exception of children and grandchildren) in the past week (0/1 scale).
Social integration: non-family | Assessed at 3 months after intervention
  This is an indicator for whether the participant talked on the phone with anyone (with the exception of children and grandchildren) in the past week (0/1 scale).
Social integration: family | Assessed at 3 weeks after intervention
  This is an indicator for whether the participant talked on the phone with children or grandchildren in the past week (0/1 scale).
Social integration: family | Assessed at 3 months after intervention
  This is an indicator for whether the participant talked on the phone with children or grandchildren in the past week (0/1 scale).
Cognitive function | Assessed at 3 weeks after intervention
  Participants will be administered the mini mental state exam, scored on a 0-11 scale, rescaled to a 0-1 scale.
Cognitive function | Assessed at 3 months after intervention
  Participants will be administered the mini mental state exam, scored on a 0-11 scale, rescaled to a 0-1 scale.
Consumption | Assessed at 3 weeks after intervention
  Participants will be asked, for the last week, amount spent on different food items (rice, wheat, pulses, milk, spices, sugar, oil, meats, vegetables, fruits, packaged foods), medical expenses, fuel, clothing, footwear, toiletries, transportation, gifts, jewelry, and other expenses.
Consumption | Assessed at 3 months after intervention
  Participants will be asked, for the last week, amount spent on different food items (rice, wheat, pulses, milk, spices, sugar, oil, meats, vegetables, fruits, packaged foods), medical expenses, fuel, clothing, footwear, toiletries, transportation, gifts, jewelry, and other expenses.
Health | Assessed at 3 weeks after intervention
  This is a 16-point score comprised of indicators for whether the respondent faced health issues in the last week, according to the question, Did you face any health issues in the past week?, and then a follow-up in which the participant specified which health issues they faced. For each of the following (unprompted) issues they faced, one point was added to their score: cold/runny nose/cough/sore throat, fever, diabetes/hypertension, excessive fatigue, dizziness, earache, chills/shivering, diarrhoea, vomiting, bloody stool/urine, body/joint pain, fall/injury, acute emergency, breathlessness, vision/hearing/skin problems, other. Those who reported no health issues were given a score of zero.
Health | Assessed at 3 months after intervention
  This is a 16-point score comprised of indicators for whether the respondent faced health issues in the last week, according to the question, Did you face any health issues in the past week?, and then a follow-up in which the participant specified which health issues they faced. For each of the following (unprompted) issues they faced, one point was added to their score: cold/runny nose/cough/sore throat, fever, diabetes/hypertension, excessive fatigue, dizziness, earache, chills/shivering, diarrhoea, vomiting, bloody stool/urine, body/joint pain, fall/injury, acute emergency, breathlessness, vision/hearing/skin problems, other. Those who reported no health issues were given a score of zero.

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL SA at IFMR, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKelway M, Banerjee A, Grela E, Schilbach F, Sequeira M, Sharma G, Vaidyanathan G, Duflo E. Effects of Cognitive Behavioral Therapy and Cash Transfers on Older Persons Living Alone in India : A Randomized Trial. Ann Intern Med. 2023 May;176(5):632-641. doi: 10.7326/M22-2496. Epub 2023 Apr 25. PMID 37094349